CLINICAL TRIAL: NCT03553992
Title: An Extended Facebook Intervention for Young Sexual and Gender Minority Smokers
Acronym: POP-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0520362; 26IR-0004 (Other Grant/Funding Number: UC Tobacco-Related Disease Research Pgm)
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Tobacco Use; Smoking; Tobacco Dependence; Tobacco Use Disorder; Tobacco Use Cessation; Tobacco Smoking; Smoking Cessation; Smoking, Cigarette; Smoking, Tobacco
Keywords: Tobacco; Gender Identity Minority; Sexual Identity Minority; Cessation; Intervention; Young Adults; Social Media; Internet; Cigarette
MeSH Terms: conditions — Tobacco Use; Smoking; Tobacco Use Disorder; Tobacco Use Cessation; Tobacco Smoking; Smoking Cessation; Cigarette Smoking | interventions — POP6 protein, S cerevisiae

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Put It Out Project (POP-6): (Experimental): a culturally tailored intervention developed for sexual and gender minority (SGM) young adults on Facebook
  Interventions: Behavioral: POP-6:
- Tobacco Status Project (TSP-6): (Experimental): the original TSP intervention (non-tailored) delivered to groups of only SGM participants on Facebook
  Interventions: Behavioral: TSP-6:

INTERVENTIONS:
Behavioral: POP-6: — 90 days of Facebook messaging, weekly live sessions targeting tobacco use and tailored to SGM young adults
  Drug: nicotine patch 14-day supply of nicotine patch
  Arms: The Put It Out Project (POP-6):
Behavioral: TSP-6: — 90 days of Facebook messaging, weekly live sessions targeting tobacco use
  Drug: nicotine patch 14-day supply of nicotine patch
  Arms: Tobacco Status Project (TSP-6):

SUMMARY:
The 2-year research plan will test the Extended Put It Out Project (POP-6) in a pilot randomized trial (N=168) compared to TSP-6, as well as comparing POP-6 and TSP-6 to the POP-3 and TSP-3 interventions from a previously-conducted trial. Participants will be young adults who smoke, identify as sexual or gender minorities (SGM), and use Facebook. Primary outcome will be biochemically verified 7-day abstinence from smoking at 3 and 6 months. Secondary outcomes will be a quit attempt (y/n), stage of change, and thoughts about tobacco abstinence at 3 and 6 months.

DETAILED DESCRIPTION:
Participants will be randomized to one of two conditions: (1) a 6-month Facebook-delivered intervention addressing tobacco use, tailored to SGM young adults; or (2) a 6-month Facebook intervention targeting tobacco use. Both interventions will include 180 days of Facebook-based messages and activities tailored to participants' readiness to quit smoking.

Assessments will occur at baseline, 3, and 6 months follow-up. Assessments will include measures on smoking, thoughts about abstinence, and SGM identity experiences. All participants who report no past 7-day smoking will be asked to give biochemical verification of smoking status with saliva nicotine test kits that will be mailed to participants.

ELIGIBILITY:
Inclusion Criteria:

* read English
* between 18 and 25 years of age
* indicate they use Facebook "most" (≥ 4) days per week
* have smoked ≥100 cigarettes in their lives and currently smoke at least 1 cigarette per day on 4 or more days of the week
* identifies as SGM
* lives in California

Exclusion Criteria:

* do not read English
* are not between 18 and 25 years of age
* indicate they do not use Facebook "most" (≥ 4) days per week
* have not smoked ≥100 cigarettes in their lives and currently smoke at least 1 cigarette per day on 4 or more days of the week
* does not identify as SGM
* does not live in California

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence at 3 months | 3 months post baseline
  Reports of no smoking in the 7 days prior to the 3 month assessment. Biochemical verification of abstinence will also be recorded.
7-day point prevalence abstinence at 6 months | 6 months post baseline
  Reports of no smoking in the 7 days prior to the 6 month assessment. Biochemical verification of abstinence will also be recorded.

SECONDARY OUTCOMES:
Reduction in cigarettes smoked by at least 50% | 3 and 6 months post baseline
  Reduction will be assessed at 3 and 6 month follow-ups
Tobacco use quit attempts | 3 and 6 months post baseline
  A Smoking Questionnaire will assess the presence and number of 24 hr quit attempts since the last assessment, used to calculate presence of at least one quit attempt (y/n) in the assessment time period. This questionnaire has good internal consistency and construct validity, and is routinely used in smoking treatment research.
Readiness to quit tobacco | 3 and 6 months post baseline
  Proportion of participants ready to quit smoking in the next month assessed at 3 and 6 months.
Thoughts About Tobacco Abstinence | 3 and 6 months post baseline
  The 4-item Thoughts About Abstinence Form, will measure thoughts about abstinence (desire to quit, abstinence self-efficacy, and perceived difficulty of quitting) on a scale from 1 ("least") to 10("most"), and abstinence goal as no goal, intermediary goal (e.g., reduced smoking), or total abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Humfleet, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Department of Psychiatry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramo DE, Thrul J, Chavez K, Delucchi KL, Prochaska JJ. Feasibility and Quit Rates of the Tobacco Status Project: A Facebook Smoking Cessation Intervention for Young Adults. J Med Internet Res. 2015 Dec 31;17(12):e291. doi: 10.2196/jmir.5209. PMID 26721211
- [Background] Thrul J, Klein AB, Ramo DE. Smoking Cessation Intervention on Facebook: Which Content Generates the Best Engagement? J Med Internet Res. 2015 Nov 11;17(11):e244. doi: 10.2196/jmir.4575. PMID 26561529
- [Background] Ramo DE, Thrul J, Delucchi KL, Ling PM, Hall SM, Prochaska JJ. The Tobacco Status Project (TSP): Study protocol for a randomized controlled trial of a Facebook smoking cessation intervention for young adults. BMC Public Health. 2015 Sep 15;15:897. doi: 10.1186/s12889-015-2217-0. PMID 26374203
- [Background] Ramo DE, Rodriguez TM, Chavez K, Sommer MJ, Prochaska JJ. Facebook Recruitment of Young Adult Smokers for a Cessation Trial: Methods, Metrics, and Lessons Learned. Internet Interv. 2014 Apr;1(2):58-64. doi: 10.1016/j.invent.2014.05.001. PMID 25045624
- [Background] Ramo DE, Liu H, Prochaska JJ. A mixed-methods study of young adults' receptivity to using Facebook for smoking cessation: if you build it, will they come? Am J Health Promot. 2015 Mar-Apr;29(4):e126-35. doi: 10.4278/ajhp.130326-QUAL-128. Epub 2014 Feb 27. PMID 24575728